CLINICAL TRIAL: NCT01579773
Title: Comparison of Body Composition & Weight Change in Users of Progestin-only Contraception During the First Year of Use
Acronym: DEXA
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 80158
Record Dates: First submitted 2012-04-10; First posted 2012-04-18 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Weight Change
MeSH Terms: conditions — Body Weight Changes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to learn if women gain weight using progestin-only methods of contraception and if so, how much. The investigators will look at users of two progestin-only methods: the levonorgestrel-containing intrauterine contraceptive (LNG-IUC) and the etonorgestrel (ENG) subdermal implant, and compare these users' weight change to that of users of a non-hormonal method, the copper intrauterine device.

The primary hypothesis is that ENG implant and LNG-IUC users' weight and body composition will increase more than the copper-IUD users. The investigators will collect body composition data using dual-energy x-ray absorptiometry (DEXA), and collect information about diet and activity using validated questionnaires.

ELIGIBILITY:
The study has finished enrolling new participants.

Inclusion Criteria:

* Participants between the ages of 18 and 45 years
* Participants starting the copper IUD or implant through their provider
* First study visit must occur within 14 days of method insertion

Exclusion Criteria:

* DMPA in the past 16 weeks
* POPs, LNG-IUC, or the implant in the past 4 weeks
* Thyroid disease
* Autoimmune disease
* Diabetes (excluding gestational)
* History of eating disorder
* Currently taking antidepressants for < 6 months
* Currently taking antipsychotics
* Currently taking oral glucocorticoids (steroids, i.e. prednisone) for more than 6 months
* Currently breastfeeding
* Less than 6 months post-partum

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants who are starting an IUD or implant through their provider could be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2010-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Weight | Baseline and 12 months
  Compare changes in body weight and BMI measurements

SECONDARY OUTCOMES:
Body composition | Baseline and 12 months
  Compare parameters including fat mass and percentage and central-to-peripheral fat ratios

CONTACTS AND LOCATIONS:
Overall Officials: Tessa E Madden, MD, MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States